CLINICAL TRIAL: NCT06224413
Title: A Postmarketing, Prospective, Multicenter, Observational, Long-Term Safety and Effectiveness Registry Study of Patients With Cerebral Adrenoleukodystrophy (CALD) Treated With Elivaldogene Autotemcel (Stargazer)
Brief Title: A Study of Participants With Cerebral Adrenoleukodystrophy (CALD) Treated With Elivaldogene Autotemcel
Acronym: Stargazer
Status: Recruiting | Type: Observational
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Other Study IDs: REG-502
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Adrenoleukodystrophy (CALD)
Keywords: Adrenoleukodystrophy; Adrenoleukodystrophy protein
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Participants with CALD treated with eli-cel in the post marketing setting will be followed in this registry study for up to 15 years after eli-cel infusion to collect real-world longitudinal data, and evaluate the outcomes.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
The main aim of this study is to assess and describe the safety outcomes, including newly diagnosed malignancies, of patients with CALD treated with eli-cel in the post-marketing setting (tradename Skysona) and to describe major functional disability (MFD)-free survival over time in participants with more advanced early active CALD. All enrolled participants with CALD treated with eli-cel in the post-marketing setting will be followed in this study for 15 years. No investigational drug product will be administered in this study. This study will enroll 120 participants with CALD treated with eli-cel in the post-marketing setting. A subpopulation of 24 participants with more advanced early active CALD will be specifically enrolled as required by the US FDA as a condition of accelerated approval and will be considered as a separate cohort for effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

Participants who fulfill the following criteria will be eligible for inclusion in this Registry Study.

* Participant must be treated with eli-cel in the post marketing setting at a center in the United States (US) that participates in the Registry Study.
* Participant must have provided an informed consent and/or assent to participate in Center for International Blood and Marrow Transplant Research (CIBMTR) registry.
* Participant must have provided an informed consent and/or assent to participate in the Registry Study.
* Participant must receive follow up care by a US-based physician with the ability to submit REG-502 data.

Registry Study Subpopulation inclusion:

Twenty-four of the 120 patients in the Registry Study must meet the following inclusion criteria which will be used to create the more advanced early active CALD subpopulation:

• Participant must meet the above inclusion criteria and have a Loes score of 4.5 through 9.0 with GdE+ (gadolinium enhancement positivity) from an MRI performed before treatment with eli-cel and with NFS of 0 or 1 at baseline.

Exclusion Criteria:

There are no exclusion criteria for this Registry Study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with CALD treated with eli-cel in the post marketing setting at a center in the US that participates in the Registry Study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2047-12-30 (Estimated); Study Completion 2047-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Each Individual Adverse Events of Interest (AEIs) | Through 15 years postinfusion
  The Sponsor considers the following events to be AEIs (which should be reported as a medically significant Serious Adverse Events [SAEs]):
  * Any newly diagnosed malignancy
  * Neutrophil engraftment failure: defined as health care provider (HCP) decision to administer back-up cells or subsequent hematopoietic stem cell transplantation (HSCT) due to neutrophil recovery failure
  * Newly acquired HIV-1 or HIV-2 infection
  * Any newly diagnosed autoimmune disorders
  * Opportunistic infections
  * Grade 3 or higher cytopenias occurring more than 60 days after eli-cel infusion
Number of Participants with Newly Diagnosed Malignancies | Through 15 years postinfusion
Number of Participants with Insertional Oncogenesis | Through 15 years postinfusion
Major Functional Disability (MFD)-Free Survival | Through 15 years postinfusion
  MFD-free survival is defined as time from drug product infusion to either a rescue cell administration or second transplant, MFD, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Through 15 years postinfusion
Number of Participants with Serious Adverse Events (SAEs) | Through 15 years postinfusion
Number of Participants with Eli-cel Related AEs | Through 15 years postinfusion
Number of Participants with Presence of Insertional Oncogenesis in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion
Number of Participants with Complete Remission in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion
Relapse-free Survival in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion
Overall Survival in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion
Number of Participants with Clinically Significant Abnormalities by Karyotyping in Bone Marrow Aspirate in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion
Number of Participants with Clinically Significant Abnormalities on Fluorescence In-situ Hybridization (FISH) and Next Generation Sequencing (NGS) in Subpopulation with Newly Diagnosed Hematologic Malignancy | Through 15 years postinfusion

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Bhirangi, MD, Study Director — bluebird bio, Inc.
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency and appropriately de-identified patient-level datasets and supporting documents may be shared (if contractually or otherwise legally permitted ) following completion of this study, submission of all applicable regulatory submissions and consistent with criteria established by bluebird bio, our collaborators (CIBMTR) and/or industry best practices to protect confidential information and maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.